CLINICAL TRIAL: NCT03625882
Title: VPRIV Drug Use-Result Survey (Japan)
Brief Title: Survey Study for Velaglucerase Alfa (VPRIV) in Japan
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: SHP-GCB-401
Record Dates: First submitted 2018-08-08; First posted 2018-08-10 (Actual); Results first posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-11

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gaucher Disease Participants Treated With VPRIV: Participants with Gaucher disease will be enrolled in this survey, who are in VPRIV treatment-naïve therapy or have been switched from another therapeutic agent for Gaucher disease.

SUMMARY:
The objective of this post-marketing survey study is to collect data to determine the safety and efficacy of velaglucerase alfa (VPRIV) in participants with Gaucher disease who are new to therapy or have been switched from another therapeutic agent for Gaucher disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants with a confirmed diagnosis of Gaucher disease
* Participants who are either naïve to treatment or participants that have been treated with another therapeutic agent for Gaucher disease
* Participants who start VPRIV treatment or transition from VPRIV clinical studies during the enrollment period

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with confirmed Gaucher disease (types 1, 2, or 3) irrespective of any age or gender who are either naïve to treatment or participants that have been treated with another therapeutic agent for Gaucher disease.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2014-09-02 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (31):
- Japan (31):
  - Konan, Kōnan, Aichi-ken
  - Nagoya, Nagoya, Aichi-ken
  - Kitakyushu, Kitakyushu, Fukuoka
  - Kurume, Kurume, Fukuoka
  - Fukuyama, Fukuyama, Hiroshima
  - Higashihiroshima, Higashihiroshima, Hiroshima
  - Obihiro, Obihiro, Hokkaido
  - Sagamihara, Sagamihara, Kanagawa
  - Sendai, Sendai, Miyagi
  - Suita, Suita, Osaka
  - Tondabayashi, Tondabayashi, Osaka
  - Kawagoe, Kawagoe, Saitama
  - Tokorozawa, Tokorozawa, Saitama
  - Moriyama, Moriyama, Shiga
  - Otsu, Ōtsu, Shiga
  - Matsue, Matsue, Shimane
  - Hamamatsu, Hamamatsu, Shizuoka
  - Iwata, Iwata, Shizuoka
  - Minato, Minato, Tokyo
  - Sumida-ku, Sumida-ku, Tokyo
  - Yonago, Yonago, Tottori
  - Chiba, Chiba
  - Gifu, Gifu
  - Hiroshima, Hiroshima
  - Kagoshima, Kagoshima
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Okayama, Okayama
  - Osaka, Osaka
  - Saitama, Saitama
  - Shizuoka, Shizuoka

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Sagara R, Ishigaki M, Otsuka M, Murayama K, Ida H, Fernandez J. Long-term safety and effectiveness of velaglucerase alfa in Gaucher disease: 6-year interim analysis of a post-marketing surveillance in Japan. Orphanet J Rare Dis. 2021 Dec 4;16(1):502. doi: 10.1186/s13023-021-02119-2. PMID 34863216
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fe94db2bf003ab47b4e

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 45 investigative sites in Japan, from 2 Sep 2014 to 14 May 2024.
Pre-assignment Details: Participants with Gaucher disease who received Recombinant Velaglucerase Alfa were enrolled. Participants received VPRIV intravenous infusion as part of a routine medical care.
Groups:
- Recombinant Velaglucerase Alfa Intravenous Infusion: Participants with Gaucher disease received Recombinant Velaglucerase Alfa intravenous infusion as part of a routine medical care.
Period: Overall Study
Arm/Group | Recombinant Velaglucerase Alfa Intravenous Infusion
Started | 63
Completed | 60
Not Completed | 3
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Arm/Group | Recombinant Velaglucerase Alfa Intravenous Infusion
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 19.8 (21.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAE) Following Initiation of Treatment With Velaglucerase Alfa
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any event that results in: death; life-threatening; requires inpatient hospitalisation or results in prolongation of existing hospitalisation; persistent or significant disability/incapacity; a congenital anomaly/birth defect or a medically important event.
Time Frame: Baseline up to end of the study (8 years)
Population: Safety Analysis Set, The safety analysis set was defined as all participants who received at least one dose of Recombinant Velaglucerase Alfa intravenous infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Velaglucerase Alfa Intravenous Infusion
Number analyzed (Participants) | 60
Participants
  Adverse Events | 42
  Serious Adverse Events | 27

2. Secondary Outcome: Number of Participants of Efficacy Categories in Assessment of Change From Baseline in Hemoglobin Concentration
Description: Number of participants of efficacy categories in assessment of change from baseline in hemoglobin concentration during the study was reported. The efficacy categories were classified as Good: increased by at least 1.5g/dL, Moderate response: increase of at least 0.5 g/dL and less than 1.5 g/dL, and Ineffective: increase less than 0.5 g/dL.
Time Frame: Baseline, Every 12 weeks up to 8 years
Population: Efficacy Analysis Set: all participants who received at least one dose of Recombinant Velaglucerase Alfa intravenous infusion. The number analyzed was the number of participants what the data was available in this outcome measure during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Velaglucerase Alfa Intravenous Infusion
Number analyzed (Participants) | 35
Participants
  Good | 11
  Moderate response | 4
  Ineffective | 20

3. Secondary Outcome: Number of Participants of Efficacy Categories in Assessment of Change From Baseline in Platelet Counts
Description: Number of participants of efficacy categories in assessment of change from baseline in platelet counts during the study was reported. The efficacy categories were classified as Good: increase of at least 30 × 10^9/L, Moderate response: increase of at least 15 × 10^9/L and less than 30 × 10^9/L, and Ineffective: less than 15 × 10^9/L.
Time Frame: Baseline, Every 12 weeks up to 8 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Velaglucerase Alfa Intravenous Infusion
Number analyzed (Participants) | 19
Participants
  Good | 9
  Moderate response | 6
  Ineffective | 4

4. Secondary Outcome: Number of Participants of Efficacy Categories in Assessment of Change From Baseline in Liver Volumes
Description: Number of participants of efficacy categories in assessment of change from baseline in liver volumes during the study was reported. The efficacy categories were classified as Good: reduction of at least 30%, Moderate response: reduction of at least 10% and less than 30%, and Ineffective: less than 10% reduction.
Time Frame: Baseline, Every 24 weeks up to 8 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Velaglucerase Alfa Intravenous Infusion
Number analyzed (Participants) | 7
Participants
  Good | 0
  Moderate response | 1
  Ineffective | 6

5. Secondary Outcome: Number of Participants of Efficacy Categories in Assessment of Change From Baseline in Spleen Volumes
Description: Number of participants of efficacy categories in assessment of change from baseline in spleen volumes during the study was reported. The efficacy categories were classified as Good: reduction of at least 30%, Moderate response: reduction of at least 10% and less than 30%, and Ineffective: less than 10% reduction.
Time Frame: Baseline, Every 24 weeks up to 8 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Velaglucerase Alfa Intravenous Infusion
Number analyzed (Participants) | 8
Participants
  Good | 3
  Moderate response | 2
  Ineffective | 3

6. Secondary Outcome: Lumbar Spine Bone Mineral Density (BMD) T-scores and Femur Neck BMD T-scores at Baseline and the Last Data Collection
Description: T-scores were the number of standard deviations (SDs) above or below the average for a young adult at peak BMD. A T-score of 0 was equal to the mean. Negative numbers indicated values lower than the mean and positive numbers indicated values higher than the mean. The reported data in this outcome measure was lumbar spine BMD T-scores and femur neck BMD T-scores related to bone density at baseline and the last data collection.
Time Frame: Baseline, at the time of last data collection (up to 8 years)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Recombinant Velaglucerase Alfa Intravenous Infusion
Number analyzed (Participants) | 1
T-score
  Lumbar Spine BMD T-scores: Baseline | -4.30 (NA) — The standard deviation was not evaluable due to low number of participants with events.
  Lumbar Spine BMD T-scores: At the last data collection | -0.30 (NA) — The standard deviation was not evaluable due to low number of participants with events.
  Femur Neck BMD T-scores: Baseline | -2.90 (NA) — The standard deviation was not evaluable due to low number of participants with events.
  Femur Neck BMD T-scores: At the last data collection | -0.60 (NA) — The standard deviation was not evaluable due to low number of participants with events.

7. Secondary Outcome: Lumbar Spine BMD Z-scores and Femur Neck BMD Z-scores at Baseline and the Last Data Collection
Description: Z-scores express the BMD as the number of SDs above or below the average BMD of a healthy participant of the same age and gender. A Z-score of 0 was equal to the mean. Negative numbers indicated values lower than the mean and positive numbers indicated values higher than the mean. The reported data in this outcome measure was lumbar spine BMD Z-scores and femur neck BMD Z-scores related to bone density at baseline and the last data collection.
Time Frame: Baseline, at the time of last data collection (up to 8 years)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Recombinant Velaglucerase Alfa Intravenous Infusion
Number analyzed (Participants) | 2
Z-score
  Lumbar Spine BMD Z-scores: Baseline: number analyzed (Participants) | 1
  Lumbar Spine BMD Z-scores: Baseline | -2.20 (NA) — The standard deviation was not evaluable due to low number of participants with events.
  Lumbar Spine BMD Z-scores: At the last data collection | -1.15 (1.202)
  Femur Neck BMD Z-scores: Baseline: number analyzed (Participants) | 1
  Femur Neck BMD Z-scores: Baseline | -0.60 (NA) — The standard deviation was not evaluable due to low number of participants with events.
  Femur Neck BMD Z-scores: At the last data collection: number analyzed (Participants) | 1
  Femur Neck BMD Z-scores: At the last data collection | -0.50 (NA) — The standard deviation was not evaluable due to low number of participants with events.

8. Secondary Outcome: Lumbar Spine BMD and Femur Neck BMD at Baseline and the Last Data Collection
Description: The reported data in this outcome measure was lumbar spine BMD and femur neck BMD related to bone density at baseline and the last data collection.
Time Frame: Baseline, at the time of last data collection (up to 8 years)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: gram per square centimeter
Arm/Group | Recombinant Velaglucerase Alfa Intravenous Infusion
Number analyzed (Participants) | 2
gram per square centimeter
  Lumbar Spine BMD: Baseline | 0.7215 (0.19304)
  Lumbar Spine BMD: At the last data collection: number analyzed (Participants) | 1
  Lumbar Spine BMD: At the last data collection | 0.3550 (NA) — The standard deviation was not evaluable due to low number of participants with events.
  Femur Neck BMD: Baseline | 0.6335 (0.11809)
  Femur Neck BMD: At the last data collection: number analyzed (Participants) | 1
  Femur Neck BMD: At the last data collection | 0.3400 (NA) — The standard deviation was not evaluable due to low number of participants with events.

9. Secondary Outcome: Number of Participants With Positive Anti-velaglucerase Alfa Antibody Test Results
Description: Number of participants with positive anti-velaglucerase alfa antibody test results was reported.
Time Frame: Baseline up to end of the study (8 years)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Velaglucerase Alfa Intravenous Infusion
Number analyzed (Participants) | 15
Participants | 2

10. Secondary Outcome: Number of Participants With Adverse Drug Reaction and Serious Adverse Drug Reaction Following Initiation of Treatment With Velaglucerase Alfa
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any event that results in: death; life-threatening; requires inpatient hospitalisation or results in prolongation of existing hospitalisation; persistent or significant disability/incapacity; a congenital anomaly/birth defect or a medically important event. Adverse drug reaction refers to AE related to administered drug.
Time Frame: Baseline up to end of the study (8 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Velaglucerase Alfa Intravenous Infusion
Number analyzed (Participants) | 60
Participants
  Adverse Drug Reaction | 14
  Serious Adverse Drug Reaction | 5

11. Secondary Outcome: Number of Participants With Adverse Reactions Categorized as Infusion Reactions Following Initiation of Treatment With Velaglucerase Alfa
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Adverse drug reaction refers to AE related to administered drug. Infusion reactions were defined as reactions occurring up to 24 hours after the start of the infusion.
Time Frame: Baseline up to end of the study (8 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Velaglucerase Alfa Intravenous Infusion
Number analyzed (Participants) | 60
Participants | 6

ADVERSE EVENTS:
Time Frame: Baseline up to end of the study (8 years)
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the survey treatment.
Arm/Group | Recombinant Velaglucerase Alfa Intravenous Infusion
All-Cause Mortality (participants affected / at risk) | 14/60
Serious Adverse Events (participants affected / at risk) | 27/60
Other Adverse Events (participants affected / at risk) | 32/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Recombinant Velaglucerase Alfa Intravenous Infusion (N=60)
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Pneumonia aspiration (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Staphylococcal sepsis (Infections and infestations) | 1
Device related sepsis (Infections and infestations) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Autoimmune neutropenia (Blood and lymphatic system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Eating disorder (Psychiatric disorders) | 1
Tension (Psychiatric disorders) | 1
Bipolar disorder (Psychiatric disorders) | 1
Myoclonus (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Myoclonic epilepsy (Nervous system disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Central sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gastroenteritis eosinophilic (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Vesicoureteric reflux (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Death (General disorders) | 1 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Pyrexia (General disorders) | 1
General physical health deterioration (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Foreign body in throat (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Recombinant Velaglucerase Alfa Intravenous Infusion (N=60)
Bronchitis (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 4
Anaemia (Blood and lymphatic system disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 3
Zinc deficiency (Metabolism and nutrition disorders) | 3
Insomnia (Psychiatric disorders) | 3
Myoclonus (Nervous system disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Hepatic function abnormal (Hepatobiliary disorders) | 6
Pyrexia (General disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT03625882/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT03625882/SAP_001.pdf